CLINICAL TRIAL: NCT03197597
Title: EUpertstrain 4 Study of Bordetella Pertussis Isolates
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Collaborators: GlaxoSmithKline (Industry); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Qiushui He, Professor, University of Turku
Other Study IDs: EUpert IV
Record Dates: First submitted 2017-06-13; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Bordetella Pertussis, Whooping Cough
Keywords: B. pertussis; Acellular vaccination; Strain variation
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Collection of nasopharyngeal swabs from the human nasopharynx. From the swab, B. pertussis bacteria is isolated and cultured and DNA is studied. However, no human DNA is used in the measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Strain isolation from the nasopharynx: A group of culture positive whooping cough patients.
  Interventions: Other: Strain isolation from the nasopharynx

INTERVENTIONS:
Other: Strain isolation from the nasopharynx — B. pertussis strains has been collected from the nasopharynx of the patients during the clinical visit

SUMMARY:
This study focus on the genetic changes of B. pertussis clinical isolates. For this panels of B. pertussis isolates has been collected during four periods in different European countries.

DETAILED DESCRIPTION:
B. pertussis is considered as a monomorphic pathogen. However, genetic changes have been observed in several antigens (pertussis toxin, pertactin, filamentous haemagglutinin and fimbriae) included in the current acellular pertussis vaccines between vaccine strains and circulating isolates.

To study genetic changes in the B. pertussis populations in Europe, four distinct panels have been collected: EUpert I in 1999-2001 including 102 isolates, EUpert II in 2004-2005 including 154 isolates, EUpert III in 2007-2009 including 140 isolates and EUpert IV in 2012-2015 including 265 isolates. Selection criteria have remained unchanged for all four collections, which enables the opportunity to study changes in B. pertussis populations during the last 15 years.

ELIGIBILITY:
Inclusion Criteria:

* B. pertussis clinical isolates should be collected from subjects from different regions and be epidemiologically unrelated.
* An equal number of isolates from vaccinated and unvaccinated subjects should be collected. Optimally, the isolates are preferred to be selected from individuals less than 5 years of age.
* For countries with large numbers of isolates in their collections, isolates should be randomly selected according to criteria above.

Exclusion Criteria:

* There is no strict exclusion criteria for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population consists of pertussis culture positive patients from nine European countries. From this population, B. pertussis clinical isolates are collected and studied.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Vaccine antigen deficient (VAD) B. pertussis clinical isolates | 24 months
  We screened a panel of 265 B. pertussis clinical isolates collected from 9 European countries. We used previously developed ELISA to measure the antigen expression of pertussis toxin (PT), filamentous haemagglutinin (FHA), pertactin (PRN) and fimbriae 2&3 (Fim2&3). In addition, we used sequencing to further characterize the pertactin gene of the bacteria.
Study of genetic changes in the B. pertussis genomic content measured by specific molecular methods | 24 months
  We studied genetic changes in the main virulence genes of B. pertussis. We genotyped pertussis toxin promoter (ptxP), pertactin (PRN), fimbriae3 (Fim3) and pertussis toxin subunit A (ptxA). Serotyping of Fimbriae (Fim), Pulsed-Field Gel Electrophoresis (PFGE) and Multiple-Locus Variable number tandem repeat Analysis (MLVA) were used for further genomic analysis.
Association between vaccine antigen deficient (VAD) B. pertussis clinical isolates and their association to the introduction of acellular pertussis vaccination (ACV) | 24 months
  We studied the association between the frequency of VAD B. pertussis clinical isolates and their association to the introduction of ACV. Data of vaccination schedules by country and number of VAD isolates were collected and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Qiushui He, MD, PhD, Principal Investigator — University of Turku
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Advani A, Hallander HO, Dalby T, Krogfelt KA, Guiso N, Njamkepo E, von Konnig CH, Riffelmann M, Mooi FR, Sandven P, Lutynska A, Fry NK, Mertsola J, He Q. Pulsed-field gel electrophoresis analysis of Bordetella pertussis isolates circulating in Europe from 1998 to 2009. J Clin Microbiol. 2013 Feb;51(2):422-8. doi: 10.1128/JCM.02036-12. Epub 2012 Nov 21. PMID 23175253
- [Background] Bouchez V, Brun D, Cantinelli T, Dore G, Njamkepo E, Guiso N. First report and detailed characterization of B. pertussis isolates not expressing Pertussis Toxin or Pertactin. Vaccine. 2009 Oct 9;27(43):6034-41. doi: 10.1016/j.vaccine.2009.07.074. Epub 2009 Aug 8. PMID 19666155
- [Background] Barkoff AM, Mertsola J, Guillot S, Guiso N, Berbers G, He Q. Appearance of Bordetella pertussis strains not expressing the vaccine antigen pertactin in Finland. Clin Vaccine Immunol. 2012 Oct;19(10):1703-4. doi: 10.1128/CVI.00367-12. Epub 2012 Aug 22. No abstract available. PMID 22914363
- [Background] Mooi FR, van Loo IH, van Gent M, He Q, Bart MJ, Heuvelman KJ, de Greeff SC, Diavatopoulos D, Teunis P, Nagelkerke N, Mertsola J. Bordetella pertussis strains with increased toxin production associated with pertussis resurgence. Emerg Infect Dis. 2009 Aug;15(8):1206-13. doi: 10.3201/eid1508.081511. PMID 19751581
- [Background] Barkoff AM, Guiso N, Guillot S, Xing D, Markey K, Berbers G, Mertsola J, He Q. A rapid ELISA-based method for screening Bordetella pertussis strain production of antigens included in current acellular pertussis vaccines. J Immunol Methods. 2014 Jun;408:142-8. doi: 10.1016/j.jim.2014.06.001. Epub 2014 Jun 10. PMID 24925807
- [Background] Caro V, Njamkepo E, Van Amersfoorth SC, Mooi FR, Advani A, Hallander HO, He Q, Mertsola J, Riffelmann M, Vahrenholz C, Von Konig CH, Guiso N. Pulsed-field gel electrophoresis analysis of Bordetella pertussis populations in various European countries with different vaccine policies. Microbes Infect. 2005 Jun;7(7-8):976-82. doi: 10.1016/j.micinf.2005.04.005. PMID 15994109
- [Background] Heikkinen E, Xing DK, Olander RM, Hytonen J, Viljanen MK, Mertsola J, He Q. Bordetella pertussis isolates in Finland: serotype and fimbrial expression. BMC Microbiol. 2008 Sep 25;8:162. doi: 10.1186/1471-2180-8-162. PMID 18816412
- [Background] van Amersfoorth SC, Schouls LM, van der Heide HG, Advani A, Hallander HO, Bondeson K, von Konig CH, Riffelmann M, Vahrenholz C, Guiso N, Caro V, Njamkepo E, He Q, Mertsola J, Mooi FR. Analysis of Bordetella pertussis populations in European countries with different vaccination policies. J Clin Microbiol. 2005 Jun;43(6):2837-43. doi: 10.1128/JCM.43.6.2837-2843.2005. PMID 15956406